CLINICAL TRIAL: NCT01513499
Title: Effect of Intranasal Oxytocin on Appetite and Caloric Intake in Humans
Brief Title: Effect of Intranasal Oxytocin on Appetite and Caloric Intake in Men and Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Austen Lawson, Assistant in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MGH1004
Record Dates: First submitted 2012-01-11; First posted 2012-01-20 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Eating Behavior
Keywords: Eating behavior; Appetite; Oxytocin; Neuropeptide
MeSH Terms: conditions — Feeding Behavior | interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator): Intranasal oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Intranasal placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal oxytocin 24 IU single-dose administration
  Other Names: Syntocinon (Novartis)
  Arms: Oxytocin
Drug: Placebo — Intranasal Placebo single-dose administration
  Arms: Placebo

SUMMARY:
Exciting advances have led to the concept that hormones can modulate appetite and food intake. Oxytocin is a peptide hormone that is released in regions throughout the brain, including areas involved in food motivation. Animal studies suggest that oxytocin may reduce food intake. The effects of oxytocin administration on eating behavior in humans, which could have important implications in eating-related disorders ranging from obesity to anorexia nervosa, have not been investigated. This double-blind placebo-controlled cross-over study of single-dose oxytocin administration investigates whether:

1. Caloric intake will decrease following administration of oxytocin versus placebo
2. Appetite will decrease following administration of oxytocin versus placebo
3. Resting energy expenditure will increase following administration of oxytocin versus placebo

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* BMI 18.5-24.9, 25-40
* Regular breakfast eater (at least 4 times per week)
* Stable weight within the past three months

Exclusion Criteria:

* Psychiatric disease
* Use of psychotropic medications
* History of eating disorder
* History of excessive exercise within the last three months
* History of diabetes mellitus
* Active substance abuse
* Hematocrit below normal range
* Gastrointestinal tract surgery (including gastrectomy, gastric bypass surgery, and small or large bowel resection)
* History of cardiovascular disease (such as hypertrophic cardiomyopathy, valvular heart disease, coronary heart disease, or coronary artery spasms)
* Untreated thyroid disease
* Tobacco use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Caloric intake | +60 minutes after drug/placebo

SECONDARY OUTCOMES:
Appetite | +55 (fasting) and +90 minutes (post-prandial) after drug/placebo
  Assessed using a Visual Analogue Scale
Resting energy expenditure | +30 minutes after drug/placebo
  Assessed using metabolic cart

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided